CLINICAL TRIAL: NCT01412944
Title: A Randomized, Double-blind, Double Dummy, Multicenter Study to Assess the Safety, Tolerability and Long-term Efficacy of Intravenous (10mg/kg) and Subcutaneous (300mg) Secukinumab in Subjects With Moderate to Severe Chronic Plaque-type Psoriasis Who Are Partial Responders to Secukinumab
Brief Title: Efficacy and Safety of Intravenous and Subcutaneous Secukinumab in Moderate to Severe Chronic Plaque-type Psoriasis
Acronym: STATURE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAIN457A2307; 2011-002510-36 (EudraCT Number)
Record Dates: First submitted 2011-08-05; First posted 2011-08-09 (Estimated); Results first posted 2015-03-18 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Plaque-type Psoriasis
Keywords: Psoriasis; plaque; inflammatory skin disease; scaly patches; AIN457; secukinumab; Moderate to severe
MeSH Terms: conditions — Psoriasis; Plaque, Amyloid; Dermatitis | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- AIN457 subcutaneous (s.c.) (Experimental): During the intravenous (I.V.) period, participants received two 150 mg s.c. injections of AIN457 at randomization and week 4, and AIN457 placebo I.V. at randomization, week 2 and week 4. During the maintenance period, participants received 300 mg s.c. of open-label AIN457.
  Interventions: Drug: secukinumab 150mg
- AIN457 I.V. (Experimental): During the I.V. period, participants received AIN457 10mg/kg I.V. at randomization, week 2 and week 4, and AIN457 placebo s.c. at randomization and week 4. During the maintenance period, participants received 300 mg s.c. of open-label AIN457.
  Interventions: Drug: secukinumab 10mg/kg i.v. regimen

INTERVENTIONS:
Drug: secukinumab 150mg — secukinumab 150mg (2 injections per dose)
  Arms: AIN457 subcutaneous (s.c.)
Drug: secukinumab 10mg/kg i.v. regimen — secukinumab 10mg/kg i.v. regimen
  Arms: AIN457 I.V.

SUMMARY:
The study will assess the safety and efficacy of intravenous (10mg/kg) and subcutaneous (300mg) secukinumab in moderate to severe chronic plaque-type psoriasis who are partial responders to secukinumab.

ELIGIBILITY:
Inclusion criteria:

* Written Informed Consent must be obtained before any assessment is performed,
* Subject must be able to understand and communicate with the investigator and comply with the requirements of the study.
* Subjects must have participated in the study CAIN457A2304 and have achieved a partial response after twelve weeks of treatment with no major protocol deviations.

A partial response is defined as having achieved ≥ PASI 50 but < 75 response.

Exclusion criteria

* Pregnant women or lactating women
* Forms of psoriasis other than chronic plaque -type
* Ongoing use of prohibited psoriasis treatments
* Ongoing use of other non-psoriasis prohibited treatments
* Previous exposure to any biologic drug directly targeting IL-17 or the IL-17 receptor, except secukinumab in study CAIN457A2304
* Active ongoing inflammation diseases other than psoriasis that might confound the evaluation of the benefits of secukinumab therapy
* UV therapy or excessive exposure to sunlight

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2011-12; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (27):
- United States (6):
  - Novartis Investigative Site, Jacksonville, Florida
  - Novartis Investigative Site, West Palm Beach, Florida
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Greensboro, North Carolina
  - Novartis Investigative Site, Greer, South Carolina
- Austria (3):
  - Novartis Investigative Site, Wels, Austria
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Vienna
- Canada (3):
  - Novartis Investigative Site, Barrie, Ontario
  - Novartis Investigative Site, Waterloo, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- France (2):
  - Novartis Investigative Site, Toulouse, France
  - Novartis Investigative Site, Rouen
- Germany (5):
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Mainz
- India (3):
  - Novartis Investigative Site, Mangalore, Karnataka
  - Novartis Investigative Site, Nagpur, Maharashtra
  - Novartis Investigative Site, Nashik, Maharashtra
- Japan (4):
  - Novartis Investigative Site, Kisarazu, Chiba
  - Novartis Investigative Site, Hachiōji, Tokyo
  - Novartis Investigative Site, Minato-ku, Tokyo
  - Novartis Investigative Site, Shinjuku-ku, Tokyo
- Novartis Investigative Site, Košice, Slovak Republic, Slovakia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study consisted of 3 study periods: I.V. (I.V. infusion and subcutaneous (s.c.) regimens given in a double-blind fashion), Maintenance and follow-up. Participants, who were identified as partial responders at week 12 of study CAIN457A2304 (NCT01406938), were eligible to roll into CAIN457A2307.
Pre-assignment Details: Participants of the CAIN457A2304 150 mg or AIN457 300 mg treatment groups, who were partial responders at week 12 of CAIN457A2304, were randomized in a 1:1 ratio to the AIN457 300 mg s.c. or AIN457 10 mg/kg I.V. treatment groups of CAIN457A2307.
Period: IV: Per Previous CAIN457A2304 Treatment
Arm/Group | AIN457 Subcutaneous (s.c.) | AIN457 I.V. | I.V. Period: AIN457 150 mg - AIN457 300 mg s.c. | AIN457 300 mg - AIN457 300 mg s.c. | AIN457 150 mg - AIN457 10 mg/kg I.V. | AIN457 300 mg - AIN457 10 mg/kg I.V.
Started | 0 | 0 | 15 | 6 | 14 | 8
Completed | 0 | 0 | 14 | 6 | 14 | 6
Not Completed | 0 | 0 | 1 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Protocol deviation | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1
Period: IV: Per CAIN457A2307
Arm/Group | AIN457 Subcutaneous (s.c.) | AIN457 I.V. | I.V. Period: AIN457 150 mg - AIN457 300 mg s.c. | AIN457 300 mg - AIN457 300 mg s.c. | AIN457 150 mg - AIN457 10 mg/kg I.V. | AIN457 300 mg - AIN457 10 mg/kg I.V.
Started | 21 | 22 | 0 | 0 | 0 | 0
Completed | 20 | 20 | 0 | 0 | 0 | 0
Not Completed | 1 | 2 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol deviation | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0
Period: Entire: IV + Maintenance
Arm/Group | AIN457 Subcutaneous (s.c.) | AIN457 I.V. | I.V. Period: AIN457 150 mg - AIN457 300 mg s.c. | AIN457 300 mg - AIN457 300 mg s.c. | AIN457 150 mg - AIN457 10 mg/kg I.V. | AIN457 300 mg - AIN457 10 mg/kg I.V.
Started | 0 | 0 | 15 | 6 | 14 | 8
Completed | 0 | 0 | 14 | 5 | 11 | 6
Not Completed | 0 | 0 | 1 | 1 | 3 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Protocol deviation | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 1 | 0
Period: Entire: IV + Maintenance
Arm/Group | AIN457 Subcutaneous (s.c.) | AIN457 I.V. | I.V. Period: AIN457 150 mg - AIN457 300 mg s.c. | AIN457 300 mg - AIN457 300 mg s.c. | AIN457 150 mg - AIN457 10 mg/kg I.V. | AIN457 300 mg - AIN457 10 mg/kg I.V.
Started | 21 | 22 | 0 | 0 | 0 | 0
Completed | 19 | 17 | 0 | 0 | 0 | 0
Not Completed | 2 | 5 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 0 | 0 | 0 | 0
Not completed — Protocol deviation | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0
Period: Follow-up
Arm/Group | AIN457 Subcutaneous (s.c.) | AIN457 I.V. | I.V. Period: AIN457 150 mg - AIN457 300 mg s.c. | AIN457 300 mg - AIN457 300 mg s.c. | AIN457 150 mg - AIN457 10 mg/kg I.V. | AIN457 300 mg - AIN457 10 mg/kg I.V.
Started | 0 | 0 | 2 | 1 | 2 | 0
Completed | 0 | 0 | 2 | 1 | 2 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AIN457 Subcutaneous (s.c.) | AIN457 I.V. | Total
Number analyzed (Participants) | 21 | 22 | 43
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.6 (14.53) | 45.7 (12.14) | 46.6 (13.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 14
  Male | 16 | 13 | 29

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants (Who Achieved a Partial Response Defined as ≥ 50% But < 75% Improvement in Psoriasis Area and Severity Index (PASI) After 12 Weeks of Treatment in Study AIN457A2304) With 75% Improvement From Baseline in PASI
Description: PASI is a combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72(maximal disease). Body is divided into 4 areas for scoring (head, arms, trunk, legs; each area is scored by itself and scores are combined for final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, erythema, induration and desquamation; scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area* area score weight of section (head: 0.1, arms: 0.2 body: 0.3 legs: 0.4).
Time Frame: Week 8
Population: The full analysis set (FAS) population was used for this analysis. The FAS included all participants to whom treatment was assigned. Only participants from the FAS, who had week 8 values, were included in the analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | AIN457 Subcutaneous (s.c.) | AIN457 I.V.
Number analyzed (Participants) | 21 | 21
Percentage of participants | 66.7 | 90.5

2. Primary Outcome: Percentage of Participants (Who Achieved a Partial Response Defined as ≥ 50% But < 75% Improvement in PASI After 12 Weeks of Treatment in Study AIN457A2304) With Investigator's Global Assessment Model 2011 (IGA Mod 2011) 0 or 1 Response
Description: The IGA mod 2011 scale is static, i.e. it referred exclusively to the participant's disease at the time of the assessment, and did not compare with any of the participant's previous disease states at previous visits. The scores are: 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate, and 4 = severe. Treatment success was defined as achievement of IGA mod 2001 score of 0 or 1.
Time Frame: Week 8
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | AIN457 Subcutaneous (s.c.) | AIN457 I.V.
Number analyzed (Participants) | 21 | 21
Percentage of participants | 66.7 | 33.3

3. Secondary Outcome: Percentage of Participants Achieving PASI 50/75/90/100 Response or IGA 0 or 1 Response
Description: PASI is a combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72 (maximal disease). Body is divided into 4 areas for scoring (head, arms, trunk, legs; each area is scored by itself and scores are combined for final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, erythema, induration and desquamation; scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area* area score weight of section (head: 0.1, arms: 0.2 body: 0.3 legs: 0.4). PASI 50, 75, 90 and 100 were defined as participants achieving ≥ 50%, 75%, 90% or 100% improvement from baseline. The IGA mod 2011 scale is static, i.e. it referred exclusively to the participant's disease at the time of the assessment, and did not compare with any of the participant's previous disease states at previous visits. The scores are: 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate and 4 = severe.
Time Frame: Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36 and 40
Population: The full analysis set (FAS) population was used for this analysis. The FAS included all participants to whom treatment was assigned. Only participants from the FAS, who had values at a given week, were included in the analysis for that week.
Measure: Number; unit: Percentage of participants
Arm/Group | AIN457 Subcutaneous (s.c.) | AIN457 I.V.
Number analyzed (Participants) | 21 | 21
Percentage of participants
  Week 2 IGA 0/1 | 9.5 | 9.5
  Week 2 PASI 75 | 19.0 | 47.6
  Week 2 PASI 50 | 85.7 | 100.0
  Week 2 PASI 90 | 0.0 | 19.0
  Week 2 PASI 100 | 0.0 | 0.0
  Week 4 IGA 0/1 | 9.5 | 47.6
  Week 4 PASI 75 | 33.3 | 76.2
  Week 4 PASI 50 | 85.7 | 95.2
  Week 4 PASI 90 | 4.8 | 28.6
  Week 4 PASI 100 | 0.0 | 9.5
  Week 8 IGA 0/1 | 33.3 | 66.7
  Week 8 PASI 75 | 66.7 | 90.5
  Week 8 PASI 50 | 90.5 | 95.2
  Week 8 PASI 90 | 9.5 | 61.9
  Week 8 PASI 100 | 0.0 | 14.3
  Week 12 IGA 0/1 | 38.1 | 71.4
  Week 12 PASI 75 | 61.9 | 85.7
  Week 12 PASI 50 | 85.7 | 95.2
  Week 12 PASI 90 | 19.0 | 66.7
  Week 12 PASI 100 | 0.0 | 14.3
  Week 16 IGA 0/1 | 28.6 | 66.7
  Week 16 PASI 75 | 66.7 | 81.0
  Week 16 PASI 50 | 85.7 | 85.7
  Week 16 PASI 90 | 14.3 | 57.1
  Week 16 PASI 100 | 0.0 | 19.0
  Week 20 IGA 0/1 | 23.8 | 61.9
  Week 20 PASI 75 | 66.7 | 81.0
  Week 20 PASI 50 | 81.0 | 85.7
  Week 20 PASI 90 | 14.3 | 57.1
  Week 20 PASI 100 | 4.8 | 14.3
  Week 24 IGA 0/1 | 23.8 | 47.6
  Week 24 PASI 75 | 52.4 | 76.2
  Week 24 PASI 50 | 81.0 | 85.7
  Week 24 PASI 90 | 19.0 | 57.1
  Week 24 PASI 100 | 9.5 | 14.3
  Week 28 IGA 0/1 | 23.8 | 42.9
  Week 28 PASI 75 | 61.9 | 61.9
  Week 28 PASI 50 | 76.2 | 85.7
  Week 28 PASI 90 | 23.8 | 38.1
  Week 28 PASI 100 | 0.0 | 14.3
  Week 32 IGA 0/1 | 14.3 | 42.9
  Week 32 PASI 75 | 57.1 | 66.7
  Week 32 PASI 50 | 76.2 | 81.0
  Week 32 PASI 90 | 19.0 | 42.9
  Week 32 PASI 100 | 0.0 | 9.5
  Week 36 IGA 0/1 | 19.0 | 52.4
  Week 36 PASI 75 | 57.1 | 61.9
  Week 36 PASI 50 | 81.0 | 76.2
  Week 36PASI 90 | 23.8 | 47.6
  Week 36 PASI 100 | 0.0 | 9.5
  Week 40 IGA 0/1 | 28.6 | 42.9
  Week 40 PASI 75 | 47.6 | 61.9
  Week 40 PASI 50 | 85.7 | 71.4
  Week 40 PASI 90 | 23.8 | 47.6
  Week 40 PASI 100 | 0.0 | 14.3

4. Secondary Outcome: Mean Percent Change From Baseline in PASI Scores
Description: PASI is a combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72(maximal disease). Body is divided into 4 areas for scoring (head, arms, trunk, legs; each area is scored by itself and scores are combined for final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, erythema, induration and desquamation; scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area* area score weight of section (head: 0.1, arms: 0.2 body: 0.3 legs: 0.4). A negative mean percentage change indicates improvement.
Time Frame: Baseline, weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36 and 40
Population: The full analysis set (FAS) population was used for this analysis. The FAS included all participants to whom treatment was assigned. Only participants from the FAS, who had post-baseline values at the given weeks, were included in the analysis for that week.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | AIN457 Subcutaneous (s.c.) | AIN457 I.V.
Number analyzed (Participants) | 21 | 21
Percent change
  Week 2 | -65.427 (14.1732) | -74.824 (10.6180)
  Week 4 | -69.804 (14.4443) | -83.063 (10.7849)
  Week 8 | -75.422 (15.0913) | -90.980 (9.6116)
  Week 12 | -76.026 (17.0949) | -89.754 (11.1194)
  Week 16 | -75.079 (18.6092) | -89.645 (13.4471)
  Week 20 | -74.494 (20.5253) | -86.816 (19.4202)
  Week 24 | -72.703 (22.4086) | -85.803 (19.8869)
  Week 28 | -72.281 (23.4549) | -80.487 (25.7435)
  Week 32 | -71.770 (22.7398) | -79.557 (27.2634)
  Week 36 | -72.151 (21.4637) | -79.329 (27.2362)
  Week 40 | -73.663 (18.2709) | -77.416 (28.5592)

5. Secondary Outcome: Percentage of Participants in Each IGA Mod 2011 Score Category
Description: The IGA mod 2011 scale is static, i.e. it referred exclusively to the participant's disease at the time of the assessment, and did not compare with any of the participant's previous disease states at previous visits. The scores are: 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate, and 4 = severe.
Time Frame: Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36 and 40
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | AIN457 Subcutaneous (s.c.) | AIN457 I.V.
Number analyzed (Participants) | 21 | 21
Percentage of participants
  week 2 - clear | 0.0 | 0.0
  week 2 - almost clear | 9.5 | 9.5
  week 2 - mild | 57.1 | 66.7
  week 2 - moderate | 33.3 | 23.8
  week 2 - severe | 0.0 | 0.0
  week 4 - clear | 0.0 | 9.5
  week 4 - almost clear | 9.5 | 38.1
  week 4 - mild | 61.9 | 47.6
  week 4 - moderate | 28.6 | 4.8
  week 4 - severe | 0.0 | 0.0
  week 8 - clear | 0.0 | 19.0
  week 8 - almost clear | 33.3 | 47.6
  week 8 - mild | 38.1 | 23.8
  week 8 - moderate | 28.6 | 9.5
  week 8 - severe | 0.0 | 0.0
  week 12 - clear | 0.0 | 14.3
  week 12 - almost clear | 38.1 | 57.1
  week 12 - mild | 33.3 | 19.0
  week 12 - moderate | 28.6 | 9.5
  week 12 - severe | 0.0 | 0.0
  week 16 - clear | 0.0 | 19.0
  week 16 - almost clear | 28.6 | 52.4
  week 16 - mild | 42.9 | 19.0
  week 16 - moderate | 28.6 | 9.5
  week 16 - severe | 0.0 | 0.0
  week 20 - clear | 4.8 | 14.3
  week 20 - almost clear | 19.0 | 52.4
  week 20 - mild | 47.6 | 23.8
  week 20 - moderate | 28.6 | 9.5
  week 20 - severe | 0.0 | 0.0
  week 24 - clear | 9.5 | 14.3
  week 24 - almost clear | 14.3 | 38.1
  week 24 - mild | 33.3 | 28.6
  week 24 - moderate | 42.9 | 14.3
  week 24 - severe | 0.0 | 4.8
  week 28 - clear | 9.5 | 4.8
  week 28 - almost clear | 14.3 | 42.9
  week 28 - mild | 47.6 | 28.6
  week 28 - moderate | 28.6 | 23.8
  week 28 - severe | 0.0 | 0.0
  week 32 - clear | 4.8 | 4.8
  week 32 - almost clear | 9.5 | 42.9
  week 32 - mild | 47.6 | 23.8
  week 32 - moderate | 38.1 | 23.8
  week 32 - severe | 0.0 | 4.8
  week 36 - clear | 0.0 | 4.8
  week 36 - almost clear | 19.0 | 52.4
  week 36 - mild | 42.9 | 19.0
  week 36 - moderate | 38.1 | 19.0
  week 36 - severe | 0.0 | 4.8
  week 40 - clear | 0.0 | 14.3
  week 40 - almost clear | 28.6 | 33.3
  week 40 - mild | 33.3 | 23.8
  week 40 - moderate | 38.1 | 23.8
  week 40 - severe | 0.0 | 4.8

6. Secondary Outcome: Percentage of Participants Who Achieved Dermatology Life Quality Index (DLQI) of 0 or 1
Description: The DLQI is a ten item general dermatology disability index designed to assess health-related quality of life in adult participants with skin diseases such as eczema, psoriasis, acne and viral warts. It is a self-administered questionnaire which includes domains of daily activity, leisure, personal relationships, symptoms and feelings, treatment and school/work activities. Each domain has 4 response categories ranging from 0 (not at all) to 3 (very much). "Not relevant" is a valid score also and is scored as 0. The DLQI total score is a sum of all 10 responses. Scores range from 0 to 30 with higher scores indicating greater health-related quality of life impairment. A DLQI of 0 or 1 indicates no impairment or little impairment, respectively. A negative mean percentage change from baseline indicates improvement.
Time Frame: Baseline, Week 8, Week 16, Week 24, Week 32,up to Week 40
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | AIN457 Subcutaneous (s.c.) | AIN457 I.V.
Number analyzed (Participants) | 21 | 21
Percentage of participants
  Baseline | 0.0 | 4.8
  Week 8 (n=20,20) | 25.0 | 75.0
  Week 16 (n=20,20) | 40.0 | 70.0
  Week 24 (n=20,20) | 40.0 | 55.0
  Week 32 (n=20,20) | 40.0 | 55.0
  Week 40 (n=20,20) | 40.0 | 55.0

7. Secondary Outcome: Mean Percent Change From Baseline in Dermatology Life Quality Index (DLQI) Scores
Description: The DLQI is a ten item general dermatology disability index designed to assess health-related quality of life in adult participants with skin diseases such as eczema, psoriasis, acne and viral worts. It is a self-administered questionnaire which includes domains of daily activity, leisure, personal relationships, symptoms and feelings, treatment and school/work activities. Each domain has 4 response categories ranging from 0 (not at all) to 3 (very much). "Not relevant" is a valid score also and is scored as 0. The DLQI total score is a sum of all 10 responses. Scores range from 0 to 30 with higher scores indicating greater health-related quality of life impairment. A negative mean percentage change from baseline indicates improvement.
Time Frame: Baseline, weeks 8, 16, 24, 32 and 40
Population: The FAS population was used for this analysis. The FAS included all participants to whom treatment was assigned. Only participants from the FAS, who had post-baseline values at the given weeks, were included in the analysis for that week.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | AIN457 Subcutaneous (s.c.) | AIN457 I.V.
Number analyzed (Participants) | 20 | 20
Percent change
  week 8 | -67.1 (28.35) | -82.4 (31.13)
  week 16 | -68.7 (32.34) | -74.8 (42.19)
  week 24 | -66.9 (29.27) | -63.2 (42.65)
  week 32 | -65.4 (34.64) | -58.1 (53.40)
  week 40 | -74.2 (24.25) | -53.8 (56.21)

8. Secondary Outcome: Mean Percent Change From Baseline in EuroQOL 5-Dimension Health Status Questionnaire (EQ-5D) Health State Assessment (From 0 to 100)
Description: The EQ-5D is an instrument used to assess a participant's health status. The instrument includes a descriptive profile and a visual analog scale (VAS). The descriptive profile includes 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension had 3 response levels: no problems, some problems and severe problems. The VAS is a vertical scale that assesses the health status from 0 (worst possible health state) to 100 (best possible health state). This outcome measures the percent change in VAS score. Positive mean percent changes indicate improvement.
Time Frame: Baseline, weeks 8, 16, 24, 32 and 40
Population: The FAS population was used for this analysis. The FAS included all participants to whom treatment was assigned. Only participants from the FAS, who had values at a given week, were included in the analysis for that week.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | AIN457 Subcutaneous (s.c.) | AIN457 I.V.
Number analyzed (Participants) | 20 | 20
Percent change
  week 8 | 71.0 (157.11) | 73.1 (99.42)
  week 16 | 76.9 (153.63) | 57.5 (98.10)
  week 24 | 74.6 (171.69) | 45.3 (82.05)
  week 32 | 80.2 (177.33) | 40.9 (80.96)
  week 40 | 87.2 (173.59) | 41.3 (86.92)

9. Secondary Outcome: Number of Participants Who Developed Anti-secukinumab Antibodies
Description: The development of anti-secunimubab anti-bodies would decrease a participant's ability to respond to secukinumab treatment.
Time Frame: Baseline, weeks 12, 24 and 40
Population: Participants from full analysis set (FAS), who had values at baseline and post-baseline, were included in the analysis. The FAS included all participants to whom treatment was assigned.
Measure: Number; unit: Number of participants
Arm/Group | AIN457 Subcutaneous (s.c.) | AIN457 I.V.
Number analyzed (Participants) | 20 | 20
Number of participants | 0 | 0

10. Secondary Outcome: Relationship Between Response to AIN457 and Failed Response to Previous Biologic Psoriasis Therapy
Description: This outcome measure was not analyzed due to the small sample size of the study (43 participants).
Time Frame: End of study
Arm/Group | AIN457 Subcutaneous (s.c.) | AIN457 I.V.
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | I.V. Period: AIN457 150 mg - AIN457 300 mg s.c. | I.V. Period: AIN457 300 mg - AIN457 300 mg s.c. | I.V. Period: AIN457 150 mg - AIN457 10 mg/kg i.v. | I.V. Period: AIN457 300 mg - AIN457 10 mg/kg i.v. | Entire Period: AIN457 150 mg - AIN457 300 mg s.c. | Entire Period: AIN457 300 mg - AIN457 300 mg s.c. | Entire Period: AIN457 150 mg - AIN457 10 mg/kg i.v. | Entire Period: AIN457 300 mg - AIN457 10 mg/kg i.v. | Follow up: AIN457 300 mg - AIN457 300 mg s.c. | Follow-up: AIN457 300 mg - 10 mg/kg i.v. | Follow-up: AIN457 150 mg - 300 mg s.c. | Follow-up: AIN457 150 mg - 10 mg/kg i.v.
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/6 | 0/14 | 0/8 | 0/15 | 0/6 | 1/14 | 0/8 | 0/1 | 0/0 | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 7/15 | 4/6 | 5/14 | 5/8 | 10/15 | 5/6 | 12/14 | 6/8 | 1/1 | 0/0 | 0/2 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | I.V. Period: AIN457 150 mg - AIN457 300 mg s.c. (N=15) | I.V. Period: AIN457 300 mg - AIN457 300 mg s.c. (N=6) | I.V. Period: AIN457 150 mg - AIN457 10 mg/kg i.v. (N=14) | I.V. Period: AIN457 300 mg - AIN457 10 mg/kg i.v. (N=8) | Entire Period: AIN457 150 mg - AIN457 300 mg s.c. (N=15) | Entire Period: AIN457 300 mg - AIN457 300 mg s.c. (N=6) | Entire Period: AIN457 150 mg - AIN457 10 mg/kg i.v. (N=14) | Entire Period: AIN457 300 mg - AIN457 10 mg/kg i.v. (N=8) | Follow up: AIN457 300 mg - AIN457 300 mg s.c. (N=1) | Follow-up: AIN457 300 mg - 10 mg/kg i.v. (N=0) | Follow-up: AIN457 150 mg - 300 mg s.c. (N=2) | Follow-up: AIN457 150 mg - 10 mg/kg i.v. (N=2)
DERMATITIS ALLERGIC (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | I.V. Period: AIN457 150 mg - AIN457 300 mg s.c. (N=15) | I.V. Period: AIN457 300 mg - AIN457 300 mg s.c. (N=6) | I.V. Period: AIN457 150 mg - AIN457 10 mg/kg i.v. (N=14) | I.V. Period: AIN457 300 mg - AIN457 10 mg/kg i.v. (N=8) | Entire Period: AIN457 150 mg - AIN457 300 mg s.c. (N=15) | Entire Period: AIN457 300 mg - AIN457 300 mg s.c. (N=6) | Entire Period: AIN457 150 mg - AIN457 10 mg/kg i.v. (N=14) | Entire Period: AIN457 300 mg - AIN457 10 mg/kg i.v. (N=8) | Follow up: AIN457 300 mg - AIN457 300 mg s.c. (N=1) | Follow-up: AIN457 300 mg - 10 mg/kg i.v. (N=0) | Follow-up: AIN457 150 mg - 300 mg s.c. (N=2) | Follow-up: AIN457 150 mg - 10 mg/kg i.v. (N=2)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ATRIOVENTRICULAR BLOCK FIRST DEGREE (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
CONJUNCTIVITIS (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
CONJUNCTIVITIS ALLERGIC (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
EYELIDS PRURITUS (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
DIARRHOEA (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
GINGIVITIS ULCERATIVE (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
ILEAL ULCER (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
TOOTHACHE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
CHEST PAIN (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
FATIGUE (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
INJECTION SITE PAIN (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
ALLERGY TO PLANTS (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SEASONAL ALLERGY (Immune system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
BRONCHITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
BRONCHITIS BACTERIAL (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
EAR INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
FOLLICULITIS (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
HELICOBACTER INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HERPES ZOSTER (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
INFLUENZA (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
NASOPHARYNGITIS (Infections and infestations) | 2 | 1 | 1 | 1 | 3 | 1 | 3 | 2 | 0 | 0 | 0 | 0
ONYCHOMYCOSIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ORAL CANDIDIASIS (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PHARYNGITIS (Infections and infestations) | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
PHARYNGITIS STREPTOCOCCAL (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
PILONIDAL CYST (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
RHINITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
SINUSITIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
TINEA PEDIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
TONSILLITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
UPPER RESPIRATORY TRACT INFECTION BACTERIAL (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
EXCORIATION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
FALL (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
JOINT INJURY (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
LIMB INJURY (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
TOOTH FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
HAEMOGLOBIN DECREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
WEIGHT DECREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
PYOGENIC GRANULOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
SKIN PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HEADACHE (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
SCIATICA (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
TENSION HEADACHE (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ENURESIS (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
NEPHROLITHIASIS (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
PHARYNGEAL OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
DERMATITIS BULLOUS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
ECZEMA (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
INTERTRIGO (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
PRURITUS GENERALISED (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
PSORIASIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
SEBORRHOEIC DERMATITIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
SKIN FISSURES (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
SKIN LESION (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
FLUSHING (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
HYPERTENSION (Vascular disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
HYPOTENSION (Vascular disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
THROMBOPHLEBITIS (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.